CLINICAL TRIAL: NCT00531349
Title: Regional Anesthesia and Endometrial Cancer Recurrence
Acronym: ECA/R
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of study population
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Daniel I. Sessler, MD, Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-532
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
Keywords: Endometrial Cancer; Anesthesia; regional; cancer recurrence; Analgesia; opioid
MeSH Terms: conditions — Neoplasms; Endometrial Neoplasms; Agnosia | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): General anesthesia and opioid analgesia for the treatment of pain after surgery.
  Interventions: Drug: Sevoflurane
- B (Active Comparator): Regional anesthesia and analgesia (epidural) combined with deep sedation or general anesthesia.
  Interventions: Procedure: propofol general anesthesia

INTERVENTIONS:
Procedure: propofol general anesthesia — Regional analgesia combined with sedation or a propofol general anesthesia
  Other Names: propofol
  Arms: B
Drug: Sevoflurane — General anesthesia
  Arms: A

SUMMARY:
The purpose of this study is to determine whether recurrence of local and metastatic cancer after open hysterectomy for stage 1 or 2 endometrial cancer is reduced when patients receive epidural anesthesia/analgesia combined with propofol sedation rather than sevoflurane anesthesia and opioid analgesia.

DETAILED DESCRIPTION:
This is a Phase III, multi-center study of patients having open hysterectomies for endometrial cancer. Patients will be randomly assigned to 1) epidural anesthesia/analgesia with propofol sedation; or 2) general anesthesia combined with postoperative patient-controlled morphine analgesia. There will be a total (maximum) of 1700 patients enrolled over a 5 year enrollment.

All patients will be premedicated with 1-3 mg IV midazolam and 1-2 µg/kg fentanyl. Patients will be randomly assigned to epidural anesthesia & analgesia with propofol sedation or to sevoflurane general anesthesia and postoperative opioid analgesia after they have met the inclusion/exclusion criteria and consent to the study.

In patients assigned to general anesthesia and opioid analgesia (General Anesthesia Group), general anesthesia will be induced with 1-3 µg/kg fentanyl and 2-4 mg/kg propofol. Tracheal intubation will be facilitated by succinylcholine or a non-depolarizing muscle relaxant; alternatively, a supraglottic airway (such as a laryngeal mask) will be used. Additional non-depolarizing muscle relaxant will be administered as deemed necessary by the attending anesthesiologist.

Anesthesia will be maintained with sevoflurane in 80% oxygen, balance nitrogen, and fentanyl. Sevoflurane and fentanyl administration will be adjusted to maintain blood pressure and heart rate within 20% of pre-operative values. The lungs will be mechanically ventilated to maintain end-tidal PCO2 near 35 mm Hg. When surgery is complete, muscle relaxant will be antagonized, if necessary, and the trachea extubated. Post-operative analgesia will be morphine, provided as needed IV or via patient-controlled pump. The initial pump setting will be for 1 mg boluses with a 6-minute lockout period and no background infusion. Additional morphine will be provided as necessary to maintain good pain control, either as needed or by changing the pump settings. Morphine will be the first-line drug; but hydromorphone will be substituted at one-fifth the morphine dose in patients who do not tolerate morphine. When pain is adequately controlled without much morphine (usually on the second postoperative day), patients will be transitioned to acetaminophen and non-steroidal anti-inflammatory analgesics; oral opioids will also be permitted if necessary.

In the Epidural Anesthesia and Analgesia group, a T8-10 epidural catheter will be inserted using a standard technique. After negative aspiration for blood, patients will be given a test dose of 3 ml of 1.5% lidocaine and 1:200,000 epinephrine. The catheter will be re-inserted or repositioned as necessary until both aspiration and test dose are negative. Each patient will be given an additional 12-18 ml bolus of 0.5% bupivacaine or 0.5% ropivacaine to provide intraoperative analgesia. The catheter will be repositioned or reinserted as necessary if a sensory block to temperature cannot be confirmed in the surgical dermatomes. Additional 5-10 ml boluses of the same solution will be given hourly during surgery to maintain anesthesia; additional boluses will be permitted at the discretion of the attending anesthesiologist.

Postoperative epidural analgesia will be supplemented with acetaminophen and/or NSAIDs if needed, or per individual sites' routine protocol. Supplemental morphine will be provided only if pain relief is inadequate, either "as needed" or by patient-controlled infusion. As soon as practical, usually on the second postoperative day, patients will be transitioned to acetaminophen and/or non-steroidal analgesics and, if necessary, oral opioids.

ELIGIBILITY:
Inclusion Criteria:

1. Primary endometrial cancer without known extension beyond the uterus i.e., believed to be Stage 1 or 2
2. Scheduled for open abdominal hysterectomy
3. Written informed consent, including willingness to be randomized epidural anesthesia/analgesia with sedation or to sevoflurane general anesthesia and postoperative opioid analgesia

Exclusion Criteria:

1. Previous surgery for endometrial cancer
2. Any contraindication to epidural anesthesia or analgesia (including coagulopathy, abnormal anatomy)
3. Any contraindication to midazolam, propofol, sevoflurane, fentanyl, or morphine
4. Age < 18 or > 85 years old
5. ASA Physical Status ≥ 4
6. Any contraindication to epidural anesthesia and analgesia (including coagulopathy, abnormal anatomy)
7. Other cancer not believed by the attending surgeon to be in long-term remission
8. Systemic disease believed by the attending surgeon or anesthesiologist to present ≥ 25% two-year mortality

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Time to metastatic spread or local cancer recurrence | every six months throughout the study, yearly thereafter

SECONDARY OUTCOMES:
Any-cause mortality | 4.4 years, 6.0 years, 7.5 years and if needed 8.9 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I. Sessler, MD, Principal Investigator — The Cleveland Clinic; Daniel I. Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No